CLINICAL TRIAL: NCT04310657
Title: mNGS Was Applied to the Study of Pathogen Identification, Precision Medication and Efficacy Evaluation of Infected Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ruilan Wang, prof, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mNGS
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: mNGS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision therapy (Experimental)
  Interventions: Diagnostic Test: mNGS
- control (No Intervention)

INTERVENTIONS:
Diagnostic Test: mNGS — Metagenomics second generation sequencing technology
  Arms: Precision therapy

SUMMARY:
1) prospectively collected the patients with the proposed infection, confirmed the infection or excluded the infection through mNGS detection combined with traditional pathogen detection methods and clinical characteristics, compared the detection performance of mNGS and traditional methods, and explored the significance of mNGS microbial map characteristics for the diagnosis/exclusion of infection; 2) real-time dynamic monitoring of the pathogen and microecology of infected patients during the targeted drug use, and evaluation of the efficacy in combination with other indicators; 3) to explore the significance of the number of pathogen sequences before the clinical withdrawal of drugs to the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* expected length of stay in ICU was > 24 h
* suspected infected patients (PSI or CPIS, qSOFA or SIRS)

Exclusion Criteria:

* Pregnant and lactating women
* Who has not signed the informed consent
* the researchers considered that others were not suitable for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  28-day mortality